CLINICAL TRIAL: NCT00863395
Title: Recalcitrant Pruritus in Cutaneous T-Cell Lymphoma
Acronym: CTCL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0705M09523
Record Dates: First submitted 2009-02-24; First posted 2009-03-18 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Cutaneous T-Cell Lymphoma
Keywords: pruritis; itch; CTCL
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Pruritus | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Skin Biopsy (Experimental)
  Interventions: Procedure: skin biopsy

INTERVENTIONS:
Procedure: skin biopsy — Lidocaine 1% c Epinephrine for local anesthesia
  Other Names: Lidocaine

SUMMARY:
The purpose of this study is to define the mechanisms that underlie the refractory pruritus (itch) in Cutaneous T-Cell Lymphoma (CTCL).

DETAILED DESCRIPTION:
Little is known about the fundamental cause of pruritus in CTCL, however we do know the malignant CD4+ T-cells of CTCL accumulate in the epidermis and are in close proximity to the neural, immune and vascular systems that influence and regulate the biology of the skin. The close proximity of malignant CD4+ T-cells with the key mediators in the itch process could result in the pruritus experienced by patients with CTCL. To accomplish this we are collecting and examining skin biopsies for CTCL patients and healthy controls to identify itch-associated local biomarkers of the disease. In addition to these skin biopsies, we are retrospectively examining existing paraffin-embedded skin biopsy tissue blocks from CTCL patients. We are performing comparative and quantitative immunohistochemical analyses on the samples. This study will help to determine which components in the skin are potential key players in the manifestation and maintenance of recalcitrant pruritus in patients with CTCL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CTCL

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Collection of biopsies from pruritic CTCL patients, non pruritic CTCL patients and controls and analysis of a panel of itch-associated local biomarkers in an attempt to characterize and quantify the components in the skin involved. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hordinsky, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States